CLINICAL TRIAL: NCT00128882
Title: Treatment of Idiopathic Thrombocytopenic Purpura in Children With Subcutaneously Administered Anti-D
Brief Title: Treatment of Idiopathic Thrombocytopenic Purpura (ITP) With Subcutaneously Administered Anti-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Kjaersgaard, Mimi, M.D. (Individual)
Responsible Party: Mimi Kjaersgaard, MD, University of Aarhus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-2005-1; 2003179; 2612-2447
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: Idiopathic Thrombocytopenic Purpura; Treatment; Anti-D; Subcutaneous; Clinical evaluation; Platelet count; IVIG
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — RHO(D) antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Anti-D — Subcutaneous injection

SUMMARY:
The purpose of this study is to describe the effect of anti-D on symptoms and platelet count in children suffering from unexplainable low platelet counts, when anti-D is administered as an injection under the skin. The hypothesis is that the injection with anti-D under the skin is as effective as anti-D given in a vein.

DETAILED DESCRIPTION:
Background:

Idiopathic thrombocytopenic purpura (ITP) in children is considered a benign hematological disease. The incidence is approximately 50 cases a year in Denmark. Approximately 25 % will experience chronic disease. Follow up and treatment of these patients is not centralized.

The drug of choice is intravenous IgG (IVIG) for treatment of ITP. The side effects are flu-like symptoms, and in rare cases aseptic meningitis. Another option is intravenous anti-D, if the child is rhesus positive. Anti-D is primarily used in North America. The effect of Anti-D is comparable with IVIG when considering the time it takes to bring the platelet count above 50,000/μL. Anti-D also causes flu-like symptoms. Establishing an i.v. access is a disadvantage to both IVIG and anti-D. For both treatments mechanism of action is not finally described.

Subcutaneous IgG substitution therapy is used for patients suffering from agammaglobulinaemia. It is therefore known, that immunoglobulin uptake is possible after subcutaneous administration. Subcutaneous anti-D has been tried in few patients suffering from chronic thrombocytopenia with positive results.

IVIG treatment is expensive compared to anti-D. Treatment of a 20 kg child costs approximately 17,000 Dkr for IVIG and 2,500 Dkr. for anti-D.

Hypothesis:

* Subcutaneous administered anti-D is as effective as IVIG/i.v. anti-D;
* Subcutaneous administered anti-D has fewer less severe side effects than IVIG/i.v. anti-D.

Purpose:

* To document the effect of subcutaneous anti-D;
* Describe complications;
* Describe aspects of the mechanism of action.

Material and Methods:

Children are eligible if admitted to a pediatric department in Denmark for diagnosis, observation or treatment of acute or chronic ITP. Examination and diagnostic work up is similar throughout the country, but not identical. No specific tests are required for diagnosis. If treatment is indicated rhesus positive children are treated with subcutaneous anti-D. Rhesus negative children are treated according to local guidelines. Specified follow-up on all children is mandatory. For research purposes one blood sample form all children is collected, and from children, who receive medical treatment, several blood samples are collected. Analysis for changes in immunological signaling peptides will be performed with special attention to the mechanism of action of anti-D.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic thrombocytopenic purpura (ITP)

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2004-11; Primary Completion 2008-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Clinical effect evaluated on clinical score scale before and after treatment at specified intervals | day 0,1,3,6,14,30, 180,360

SECONDARY OUTCOMES:
Platelet count | day 0, 1, 3, 6, 14, 30, 180, 360

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Kjaersgaard, MD, Study Director — University of Aarhus, Clinical Institute, Department of Pediatrics; Henrik Hasle, MD PhD, Principal Investigator — Skejby Hospital, University of Aarhus, Department of Pediatrics
Locations (17):
- Denmark (17):
  - Aalborg University Hospital, Department of Pediatrics, Aalborg
  - Skejby Hospital, Aarhus University Hospital, Department of Pediatrics, Aarhus N
  - Amager Hospital, Department of Pediatrics, Copenhagen S
  - Rigshospitalet, Copenhagen University Hospital, Pediatric Clinic II, Copenhagen Ø
  - Esbjerg Hospital, Department of Pediatrics, Esbjerg
  - Gentofte Hospital, Department of Pediatrics, Gentofte Municipality
  - Herning Hospital, Department of Pediatrics, Herning
  - Hjoerring Hospital, Department of Pediatrics, Hjørring
  - Holbæk Hospital, Department of Pediatrics, Holbæk
  - Hvidovre Hospital, Department of Pediatrics, Hvidovre
  - Kolding Hospital Department of Pediatrics, Kolding
  - Nykøbing F, Department of Pediatrics, Nykøbing Falster
  - Næstved Hospital, Department of Pediatrics, Næstved
  - Odense University Hospital, Odense C
  - Randers Hospital, Department of Pediatrics, Randers
  - Sønderborg Hospital, Department of Pediatrics, Sønderborg
  - Viborg Hospital, Department of Pediatrics, Viborg